CLINICAL TRIAL: NCT03204552
Title: Dalin Tzu Chi General Hospital
Brief Title: Tzu Chi Health Study (Diabetes and Cardiometabolic Health Components)
Acronym: TCHS
Status: Completed | Type: Observational
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Tina H. T. Chiu, Nutritionist, Dalin Tzu Chi General Hospital
Other Study IDs: TCHS-01
Record Dates: First submitted 2017-06-21; First posted 2017-07-02 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Diabetes; Fatty Liver; Cardiometabolic Health; Body Mass Index
MeSH Terms: conditions — Diabetes Mellitus; Fatty Liver | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
To determine the effect of diet and lifestyle, particularly vegetarian diets on chronic degenerative disease outcomes in a cohort of Taiwanese Buddhists participants

DETAILED DESCRIPTION:
How did the study come about? The Tzu Chi Health Study (TCHS) began in 2007 with the goal of investigating the role of a vegetarian diet on health outcomes.

Founded in 1966, the Buddhist Tzu Chi Foundation is a leading humanitarian organization with a worldwide base of more than 5 million supporters and volunteers. Tzu means "compassion" and Chi means "relief". The organization has chapters in 47 countries on six continents, which carry out the missions of Charity, Medicine, Education, and Humanistic Culture, and delivered aid to 67 countries, to date. Today in Taiwan, there are six Tzu Chi hospitals: four large teaching hospitals (in Hualien, Dalin, Taipei, and Taichung), and two small community hospitals (in Kuanshan and Yuli). Tzu Chi has established in Taiwan a comprehensive educational system from pre-school to graduate school, including Tzu Chi University (housing now a leading medical school in Taiwan) and operates Da Ai (Great Love) TV, a global satellite television station that runs in part on proceeds from its on-going recycling program.

For reasons of compassion and environmental conservation, a vegetarian diet is suggested, but not required, for Tzu Chi Commissioners. This population of Commissioners is a non-smoking, non-drinking population, with a wide range of dietary practice: about 30% are vegetarians, 38% partial vegetarians, and 32% omnivores. A free comprehensive health examination is available for Tzu Chi commissioners at Tzu Chi hospitals every two years. TCHS was established at Dalin Tzu Chi Hospital, where both Commissioners and patients coming for health examinations have been invited to participate in the study.

This study provides a unique opportunity to examine the health of East Asian Vegetarians. Much evidence for the health effects of a vegetarian diet are currently from western populations, namely the Seventh Day Adventists and the British vegetarians, while there is very little evidence on East Asian vegetarians who consume a different vegetarian diet.

Who is in the sample? A total of 6002 subjects have enrolled in the study. More than 70% of the participants are Tzu Chi Commissioners. The female-to-male ratio is about 2:1.

How are the study subjects followed up? Participants are followed through several methods: (1) every three years, participants were invited back for detailed health examination. (2) Follow-up questionnaire sent to participants who did not return for health examination. (3) Linkages to the National Health Insurance Database and death registry.

What has been measured? Dietary, lifestyle and medical and family histories on diseases were obtained through a questionnaire, administered by interviewers. Biochemical and anthropometric data was collected through physical exams.

* Dietary questionnaire: A dietary questionnaire has been administered, with trained research dietitians as interviewers. The questionnaire was adopted from the National Nutrition Survey in Taiwan.
* Biochemical variables: CBC, fasting glucose, lipid profile (TCH, LDL, HDL, TG), BUN, Cr, ALT, AST, and UA. In addition, homocysteine, serum vitamin B12, folate, and C-reactive protein (CRP) are available for 1500 subjects.
* Blood: Extra blood samples have been obtained and stored for 3500 subjects and will be available for future investigation.
* Anthropometric variables: body weight, height, waist circumference, % body fat (with BIA), blood pressure, pulse wave velocity, bone mineral density through DXA (at spine for female and hip for male), lung function test (spirometric), abdominal sonography, colonoscopy, esophageal-gastro-duodenal-scopy, chest X-ray, KUB.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals who came to Dalin Tzu Chi Hospital for health examination between 2007 to 2009.
* Willing to participate in the study, be interviewed on questionnaires on demographics, diet, and lifestyle; willing to release health examination data for study purpose, and willing to be followed-up on health outcome

Exclusion Criteria:

* Participants less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: More than 70% of the participants are Tzu Chi Commissioners. The female-to-male ratio is about 2:1, and about one-third of study participants were vegetarians.
Sampling Method: Non-Probability Sample
Enrollment: 6002 (Actual)
Dates: Start 2007-10-15 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Diabetes | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 years
  Diabetes incidence as determined through biochemical markers (fasting blood sugar, HbA1C), disease follow-up questionnaire, and medical records
Fatty liver | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 years
  Fatty liver incidence as assessed through ultrasonography, disease follow-up questionnaire, and medical records
Change in cardiometabolic health markers | The above outcomes would be measured at baseline, 3rd year, and 6th year
  plasma lipids (cholesterol, triglyceride), pulse wave velocity, blood pressures; these markers may be combined to calculate metabolic syndrome or other scores representing metabolic health
Change in BMI | The above outcomes would be measured at baseline, 3rd year, and 6th year
  Change in BMI (calculated through height and weigh)

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Lon Lin, MD, Study Chair — Tzu Chi Medical Foundation
Locations (1):
- Dalin Tzu Chi Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chiu TH, Huang HY, Chen KJ, Wu YR, Chiu JP, Li YH, Chiu BC, Lin CL, Lin MN. Relative validity and reproducibility of a quantitative FFQ for assessing nutrient intakes of vegetarians in Taiwan. Public Health Nutr. 2014 Jul;17(7):1459-66. doi: 10.1017/S1368980013001560. Epub 2013 Jun 20. PMID 23782894
- [Result] Chiu TH, Huang HY, Chiu YF, Pan WH, Kao HY, Chiu JP, Lin MN, Lin CL. Taiwanese vegetarians and omnivores: dietary composition, prevalence of diabetes and IFG. PLoS One. 2014 Feb 11;9(2):e88547. doi: 10.1371/journal.pone.0088547. eCollection 2014. PMID 24523914
- [Result] Chiu THT, Pan WH, Lin MN, Lin CL. Vegetarian diet, change in dietary patterns, and diabetes risk: a prospective study. Nutr Diabetes. 2018 Mar 9;8(1):12. doi: 10.1038/s41387-018-0022-4. PMID 29549240
- [Result] Chiu TH, Lin MN, Pan WH, Chen YC, Lin CL. Vegetarian diet, food substitution, and nonalcoholic fatty liver. Tzu Chi Med J. 2018 Apr-Jun;30(2):102-109. doi: 10.4103/tcmj.tcmj_109_17. PMID 29875591